CLINICAL TRIAL: NCT01166061
Title: An Escalating, Multiple-dose Study in Grass Allergic Subjects to Assess the Safety of Intradermal Injection of ToleroMune Grass
Brief Title: Safety and Tolerability of ToleroMune Grass in Grass Allergic Subjects With Rhinoconjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry)
Responsible Party: Dr Rod Hafner, VP R&D, Circassia Ltd
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TG001
Record Dates: First submitted 2010-07-08; First posted 2010-07-20 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Allergy
Keywords: Grass Allergy; Immunotherapy; Rhinoconjunctivitis; ToleroMune Grass
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): Subjects to receive either active or placebo
  Interventions: Biological: Placebo; Biological: ToleroMune Grass
- Cohort 2 (Experimental): Subjects to receive either active or placebo comparator
  Interventions: Biological: Placebo; Biological: ToleroMune Grass
- Cohort 3 (Experimental): Subjects to receive either active or placebo comparator
  Interventions: Biological: Placebo; Biological: ToleroMune Grass
- Cohort 4 (Experimental): Subjects to receive either active or placebo comparator
  Interventions: Biological: Placebo; Biological: ToleroMune Grass
- Cohort 5 (Experimental): Subjects to receive either active or placebo comparator
  Interventions: Biological: Placebo; Biological: ToleroMune Grass

INTERVENTIONS:
Biological: Placebo — Solution resembling active solution but without peptides
Biological: ToleroMune Grass — 1 x4 administrations 4 weeks apart

SUMMARY:
Grass pollen allergens are universally recognised as a major cause of allergic diseases in humans and animals, including asthma, allergic rhinitis, conjunctivitis and dermatitis. Worldwide, at least 40% of allergic patients are sensitized to grass pollen allergens and between 50-90% of hayfever or seasonal allergy sufferers are allergic to grass pollen.

ToleroMune Grass is a novel, synthetic, allergen-derived peptide desensitising vaccine, currently being developed for the treatment of grass allergy.

The purpose of the present study is to evaluate the safety and tolerability of multiple ascending doses of ToleroMune Grass in subjects allergic to grass.

DETAILED DESCRIPTION:
This study is designed as a randomised, double-blind, placebo-controlled study to evaluate the safety and tolerability of escalating multiple doses of ToleroMune Grass in subjects with a documented history of allergic rhinoconjunctivitis on exposure to grass. The efficacy of ToleroMune HDM will also be explored LPSR, EPSR, CPT and levels of grass specific IgE.

The study will consist of 3 study periods. In Period 1, Screening will be performed up to a maximum of 6 weeks before randomisation.

Period 2 (Treatment Period) will consist of 4 visits (Visits 3A-3D) four weeks apart. The first cohort will receive the lowest dose and successive dose groups will increasing doses of ToleroMune Grass, provided the first administration of the previous dose was safe and well tolerated.

In Period 3, 2 Post-treatment Challenge visits will take place, the first will be 2 weeks after the last administration in the Treatment Period and the second will be 17 weeks after the first administration. Follow-up will be conducted 3-10 days after the second PTC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years
* Minimum 2 year history of rhinoconjunctivitis on exposure to grass
* Positive skin prick test to whole grass allergen
* LPSR to whole grass allergen 8-10 hours after intradermal injection of greater than 35mm diameter response
* Positive CPT to whole grass allergen with a score ≥4

Exclusion Criteria:

* Subjects with a history of asthma
* Subjects with an FEV1 <80% of predicted
* Subjects with a rye grass specific IgE >100 kU/L
* Subjects with an acute phase skin response to whole grass allergen with a mean wheal diameter > 50 mm
* Subjects who score >1 for redness of conjunctiva or who have any watering or itchiness in the eye before administration of the CPT
* Treatment with beta-blockers, alpha-adrenoreceptor blockers, tranquillisers or psychoactive drugs
* History of any significant disease or disorder (e.g. cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple intradermal injections of ToleroMune Grass in grass allergic subjects with allergic rhinoconjunctivitis | Upto 22 weeks

SECONDARY OUTCOMES:
Area of Late Phase Skin Response | Baseline and 14 weeks
Area of Early Phase Skin Response | Baseline and 14 weeks
Change in CPT score | Baseline and 4 weeks
Grass specific IgG4 | Baseline and 14 weeks
Change in CPT score | Baseline and 14 weeks
Area of Early Phase Skin Response | Baseline and 17 weeks
Grass specific IgE | Baseline and 17 weeks
Area of Late Phase Skin Response | Baseline and 17 weeks
Change in CPT score | 17 weeks after start of treatment
Change in CPT score | Baseline and 8 weeks
Change in CPT score | Baseline and 12 weeks
Grass specific IgE | Baseline and 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Hebert, MD, Principal Investigator — Centre de recherche appliquée en allergie de Quebec
Locations (1):
- Centre de Recherche Appliqué en Allergie de Québec, Québec, Quebec, Canada